CLINICAL TRIAL: NCT04906473
Title: A Phase Ⅰ Clinical Study of Single-arm, Open, Single/Multiple Dose Escalation and Dose Extension to Assess the Safety, Tolerability, Pharmacokinetic, Pharmacodynamics and Efficacy of KY100001 in Patients With Advanced Solid Tumors
Brief Title: Safety,Tolerability, Pharmacokinetic,Pharmacodynamics and Efficacy of KY100001 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KPC/KY100001/C101
Record Dates: First submitted 2021-05-18; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumor
Keywords: biliary duct cancer; glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: Single-arm, open, single/multiple dose escalation (100mg/d, 200mg/d, 350mg/d, 550mg/d, 750mg/d) and dose Extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KY100001 (Experimental): KY100001; Tablet; Oral route; Dose escalation and dose extension
  Interventions: Drug: KY100001

INTERVENTIONS:
Drug: KY100001 — KY100001; Tablet; Oral route; Dose escalation and dose extension

SUMMARY:
to assess the safety,tolerability, pharmacokinetic,pharmacodynamics and efficacy of KY100001 in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* 1) Participate in the study voluntarily and sign the informed consent;
* 2) 18≤ age ≤75 years old, gender is not limited;
* 3) Dose escalation stage: patients with advanced solid tumor proven histologically or cytologically without standard treatment regimen, or with recurrence or progression after standard treatment, WHO are ineffective or intolerant to standard treatment regimen (for patients with glioma, WHO grade II, III and IV can be included);
* 4) Dose expansion phase IDH1 mutation positivity in part A/B: Non-cholangiocarcinoma/glioma: Any of the following conditions are allowed: A) Subjects provide genetic test report to prove IDH1 mutation positivity (NGS or qPCR);B) Subjects who voluntarily undergo tumor biopsy and/or blood sample collection for genetic testing and the test results are positive;C) Subjects can provide the last FFPE sample or pathological slides (at least 10 consecutive white slides) and voluntarily accept blood sample collection for genetic testing, and the test result is positive;Patients with cholangiocarcinoma/glioma: Any of the following conditions are allowed: a) Subjects who provide prior genetic testing report demonstrating IDH1 mutation positivity (NGS or qPCR);B) Subjects can provide the most recent FFPE sample or pathological section (at least 10 consecutive white films) or tissue biopsy sample (patients with cholangiocarcinoma should also voluntarily accept blood sample collection) for genetic testing, and the test result is positive;
* 5) Dose Expansion Phase A: Patients with advanced solid tumors with IDH1 gene mutation positive, proven histologically or cytologically, without standard treatment regimens, or relapse or progression after standard treatment, ineffective or intolerant to standard treatment regimens;
* 6) Dose expansion phase B: patients with cholangiocarcinoma/high-grade glioma (WHO grade III &IV) with IDH1 gene mutation positive, histologically or cytologically proven, WHO do not have a standard treatment regimen, or WHO relapse or progress after standard treatment, are ineffective or intolerant to the standard treatment regimen.Cohort 1: a) Histologically proven stage II-IV cholangiocarcinoma with IDH1 gene mutation positive, not eligible for radical resection, transplantation, or ablation;B) disease progression after treatment with a fluorouracil or gemcitabine basal regimen;C) at least one measurable lesion that has not previously undergone radiotherapy, chemoembolization, radioembolization or other local ablation procedures;Cohort 2: a) high-grade gliomas with IDH1 gene mutation positivity (WHO grade III &IV);B) The number of disease progression ≤2 times during screening;C) At least one previous CEMRI + perfusion MRI;D) at least one measurable lesion ≥1cm (according to RANO criteria);
* 7) At least one measurable lesion (non-glioma according to RECIST v1.1 criteria;Brain glioma according to RANO criteria);
* 8) Dose increasing stage: non-glioma patients (Eastern Cooperative Cancer Group (ECOG) score: 0-2) glioma patients (KPS score ≥50);Dose extension stage: non-glioma patients (ECOG score: 0-1 points);Glioma patients (KPS score ≥50);
* 9) Expected survival ≥3 months;
* 10) Within 7 days prior to the administration of the study drug, laboratory tests have met the following criteria.Absolute neutrophils count (ANC) ≥ 1.5×109 /L;Platelet count ≥ 80×109 /L;Hemoglobin ≥ 90 g/L;Serum creatinine ≤ 1.5x upper normal range (ULN) or creatinine clearance rate (CRCL) ≥ 60mL/min (estimated according to Cockcroft-Gault formula);Total bilirubin ≤ 1.5 X ULN or ≤ 2 X ULN (for patients with liver metastasis);AST and ALT≤ 2.5 X ULN or ≤ 5 X ULN (for patients with liver metastasis);Alkaline phosphatase ≤ 2.5 X ULN or ≤ 5 X ULN (for patients with bone metastases and/or suspected disease related liver or bile duct involvement);International Normalized Ratio or Prothrombin Time≤ 1.3x ULN;Partial activated thromboplastin time (APTT) ≤ 1.5 X ULN;
* 11) Fertile men and women of reproductive age must agree to use reliable contraception from the time of signing the informed consent until 180 days after the last dose of the study drug.Women of childbearing age include pre-menopausal women and women within 2 years after menopause.Blood pregnancy test results of women of reproductive age must be negative no more than 7 days before the first study drug administration.

Exclusion Criteria:

* 1) Allergic constitution, or previous history of severe allergy, or known allergy to the active ingredients and excipients of the study drug;
* 2) Surgical therapy, chemotherapy, radiation therapy, immunotherapy, molecular targeted therapy, or any other anti-tumor therapy within 4 weeks prior to the first administration of the study drug;
* 3) Non-glioma patients: untreated patients with brain metastases who have symptoms or require treatment to control their symptoms;Or had used any radiation, surgical or other treatment, including treatment to control symptoms, within 2 months prior to the first administration of the study drug;Patients with glioma: Patients who received an unsteady dose of dexamethasone exceeding the equivalent dose of 5mg/ day 5 days before MRI screening;
* 4) Had any of the following heart conditions: a) Had grade III-IV heart failure according to the New York Heart Association's cardiac function rating within 28 days prior to the first administration of the study drug, or had left ventricular ejection fraction (LVEF) ≤50% in Echo within 7 days prior to the first administration of the study drug;B) The history of myocardial infarction in the previous 6 months was screened;C) known unstable angina;D) known severe or uncontrolled ventricular arrhythmias;E) Screening-phase Fridericia calibrated QT interval (QTCF) ≥450 ms (male), ≥470 ms (female), or other factors that increase the risk of prolonged QTC or arrhythmic events (such as heart failure, low potassium, and a family history of long QT syndrome);F) In the screening period, there was hypertension that was still poorly controlled after drug treatment (systolic blood pressure ≥160mmHg, diastolic blood pressure ≥ 100mmHg);
* 5) Difficulty in swallowing or suffering from gastrointestinal diseases or other malabsorption conditions that affect drug absorption, such as intestinal obstruction, Crohn's disease, ulcerative colitis, short bowel syndrome, gastric emptydisturbance;Or severe gastrointestinal related toxicity that does not recover below grade 2 prior to initial administration;Or clinically significant or acute gastrointestinal disease;
* 6) Previous interstitial pulmonary disease, pulmonary fibrosis, drug-induced interstitial pulmonary disease, or radiation pneumonia disease or history;
* 7) Evidence of severe or uncontrolled liver or kidney disease;
* 8) Hepatitis B virus infection (HBcAb positive and HBV DNA lower than the detection limit could be included);Or people infected with hepatitis C virus (defined as HCV antibody positive);Or persons infected with the human immunodeficiency virus (defined as HIV-positive);
* 9) Active severe infection requiring anti-infective treatment or unexplained fever over 38℃ within 28 days prior to the first administration of the study drug;
* 10) Prior to the initial administration of the study drug, any toxicity from prior antitumor therapy had not returned to CTCAE 5.0 grade ≤1 (except for grade 2 alopecia, which could be included in secondary peripheral neuropathy determined by the investigator and medical examiner to be primary residual toxicity or stable from prior chemotherapy);
* 11) Participated in other clinical trials within 28 days prior to the first administration of the study drug;
* 12) Use of CYP2C8, CYP3A strong inhibitor or inducer within 2 weeks before the first administration of the drug in this study;
* 13) Use of drugs known to extend the Qt /QTc interval within 2 weeks before the first administration of the study drug;
* 14) Pregnant or lactating women;
* 15) The investigator believes that there is any abnormal clinical or laboratory examination or other reasons and he/she is not suitable to participate in the clinical investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with abnormal vital signs | through study completion, an average of 12 weeks
  To evaluate the safety of KY100001 in subjects with advanced solid cancer in terms of abnormal vital signs
Number of subjects with abnormal physical examination | through study completion, an average of 12 weeks
  To evaluate the safety of KY100001 in subjects with advanced solid cancer in terms of abnormal physical examination
Number of subjects with abnormal laboratory examination | through study completion, an average of 12 weeks
  To evaluate the safety of KY100001 in subjects with advanced solid cancer in terms of abnormal laboratory examination
Number of subjects with abnormal electrocardiogram | through study completion, an average of 12 weeks
  To evaluate the safety of KY100001 in subjects with advanced solid cancer in terms of abnormal electrocardiogram
Change from baseline in ECOG score | through study completion, an average of 12 weeks
  To evaluate the safety of KY100001 in subjects with advanced solid cancer in terms of ECOG score

SECONDARY OUTCOMES:
Pharmacokinetics of KY100001: Cmax | 4 weeks
  Pharacokinetic evaluation in terms of Cmax
Pharmacokinetics of KY100001: Tmax | 4 weeks
  Pharacokinetic evaluation in terms of Tmax
Pharmacokinetics of KY100001: T1/2 | 4 weeks
  Pharacokinetic evaluation in terms of T1/2
Pharmacokinetics of KY100001: AUC | 4 weeks
  Pharacokinetic evaluation in terms of AUC
The relationship between 2-hydroxyglutaric acid (2-HG) level and curative effect | 4 weeks
  biomarker evaluation in terms of 2-hydroxyglutaric acid (2-HG)
Objective Response Rate (ORR) | through study completion, an average of 12 weeks
  effectiveness evaluation in terms of Objective Response Rate (ORR)
Overall Survival (OS) | through study completion, an average of 12 weeks
  effectiveness evaluation in terms of Overall Survival (OS)
Progression-Free Survival (PFS) | through study completion, an average of 12 weeks
  effectiveness evaluation in terms of Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, prof., Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No